CLINICAL TRIAL: NCT05489458
Title: Predictive Factors for Resection and Survival in Type A Borderline Resectable Pancreatic Ductal Adenocarcinoma Patients After Neoadjuvant Therapy: A Retrospective Cohort Study
Brief Title: Predictive Factors for Resection and Survival in Type A Borderline Resectable Pancreatic Ductal Adenocarcinoma Patients After Neoadjuvant Therapy
Acronym: PF-BARNA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: BUSQUETS, JULI (Other)
Responsible Party: Sponsor-Investigator, BUSQUETS, JULI, Principal Investigator, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Other Study IDs: HUB-BR-PDAC-2022
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: BR-PDAC; Pancreatic Ductal Adenocarcinoma; Borderline Resectable; CA 19-9; Anatomical
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exploratory Surgery with Resection: Type A BR-PDAC patients that underwent surgical exploration after neoadjuvant therapy and had their tumors resected.
  Interventions: Procedure: Resection
- Exploratory Surgery without Resection: Type A BR-PDAC patients that underwent surgical exploration after neoadjuvant therapy and did not have their tumors resected.
  Interventions: Procedure: No Resection

INTERVENTIONS:
Procedure: Resection — Type A BR-PDAC patients who had a favorable tumor/vascular structures relationship confirmed during surgical exploration underwent resection.
  Groups: Exploratory Surgery with Resection
Procedure: No Resection — Type A BR-PDAC patients who did not have a favorable tumor/vascular structures relationship confirmed during surgical exploration did not undergo resection.
  Groups: Exploratory Surgery without Resection

SUMMARY:
Radical surgical resection is the only curative treatment option for pancreatic cancer, but borderline resectable tumors have a high probability of incomplete exeresis. Although neoadjuvant therapy can improve the chances of complete exeresis, not all patients respond as expected.

DETAILED DESCRIPTION:
Pancreatic cancer is an important cause of cancer-related death worldwide. Radical surgical resection still is the only curative treatment option today, but not all tumors are considered resectable. Among resectable tumors, some are deemed borderline and have a high probability of incomplete exeresis. Neoadjuvant therapy (NAT) can be a game-changer for borderline cases, and there is a lack of evidence on the predictive factors associated with resectability after neoadjuvant treatment.

This study aims to assess the prognostic factors for resectability and survival after NAT in type A borderline resectable pancreatic ductal adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old.
* Both sexes.
* Diagnosed with a type A BR-PDAC between January 2010 and December 2019.
* Minimum follow-up period of 12 months.

Exclusion Criteria:

* Patients diagnosed with a type B or type C BR-PDAC.
* Patients diagnosed with a type A BR-PDAC who had disease progression prior to receiving NAT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All BR-PDAC patients that required an evaluation by the Digestive and General Surgery Department from January 2010 to December 2019 were assessed for eligibility. These patients live within the Bellvitge University Hospital (tertiary level hospital) service area.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
The number of type A BR-PDAC patients who, after receiving NAT (≥3 cycles), undergo resection. | From 6 weeks until the end of the observation period (December 2019) or death (whichever occurs first)
  NAT was administered up to 6 cycles, and cycles were administered every 2 weeks.
  The minimum time interval between the last NAT session and surgery was 4 weeks.
The evolution of the plasmatic levels of CA 19-9 from starting NAT until the surgical exploration. | Up to 16 weeks
  NAT was administered up to 6 cycles, and cycles were administered every 2 weeks.
  The minimum time interval between the last NAT session and surgery was 4 weeks.
The evolution of the degree of vascular involvement in 64-MDCT scans from starting NAT until the surgical exploration. | Up to 16 weeks
  We will evaluate the tumor's anatomical relationship with neighboring vascular structures before and after NAT, measured with 64-MDCT (multidetector computerized tomography) scans.
  NAT was administered up to 6 cycles, and cycles were administered every 2 weeks.
  The minimum time interval between the last NAT session and surgery was 4 weeks.
Overall survival | From starting NAT until the end of the observation period (December 2019) or death (whichever occurs first).
  Time until death (from any cause)
The evolution of the plasmatic levels of CA 19-9 | From starting NAT until end of the observation period (December 2019) or death (whichever occurs first).
The evolution of the degree of vascular involvement in 64-MDCT scans | From starting NAT until end of the observation period (December 2019) or death (whichever occurs first).
  The tumor's anatomical relationship with neighboring vascular structures; measured with 64-MDCT scans.
Progression-Free Survival | From starting NAT until end of the observation period (December 2019) or disease progression (whichever occurs first).
  Time until disease progression
The evolution of the plasmatic levels of CA 19-9 | From starting NAT until end of the observation period (December 2019) or disease progression (whichever occurs first).
The evolution of the degree of vascular involvement in 64-MDCT scans | From starting NAT until end of the observation period (December 2019) or disease progression (whichever occurs first).
  The tumor's anatomical relationship with neighboring vascular structures; measured with 64-MDCT scans.

SECONDARY OUTCOMES:
The number (percentage) of deaths at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
The number (percentage) of patients presenting disease progression at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
  Disease progression will be considered as the development of metastatic disease and/or an increase in the primary tumor size.
The number (percentage) of patients presenting stable disease at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
  Stable disease will be considered as an insufficient increase or reduction in the primary tumor size or in its relationship with neighboring vascular structures (i.e., cases that cannot be classified as responders).
The number (percentage) of patients considered responders at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
  Patients will be considered responders when the primary tumor presents a reduction in size and/or in its relationship with neighboring vascular structures.
The number (percentage) of patients surgically explored at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
The Resection Rate at the end of the observation period. | From starting NAT until end of the observation period (December 2019)
  The Resection Rate will be calculated by dividing the total number of resections performed by the total number of patients treated with NAT.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Secanella, MD, Principal Investigator — Bellvitge University Hospital

IPD SHARING:
Plan to Share IPD: Undecided